CLINICAL TRIAL: NCT05725057
Title: A Phase 2a, Proof of Concept Study Evaluating the Safety and Tolerability of AX-158 in Patients With Mild to Moderate Plaque Psoriasis
Brief Title: Proof of Concept Study of AX-158 in Patients With Mild to Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Artax Biopharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AX-158-1011
Record Dates: First submitted 2023-01-26; First posted 2023-02-13 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Prospective, randomized, multicenter, double-blind, placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AX-158 - (Arm 1) (Active Comparator): AX-158 Dosage:5 mg capsules Form: Capsule Frequency - 2 capsules daily taken orally Duration - 28 consecutive days
  Interventions: Drug: AX-158
- Placebo - (Arm 2) (Placebo Comparator): Placebo Dosage: NA Form: Capsule Frequency: 2 capsules daily taken orally Duration: 28 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AX-158 — Subjects randomized to this arm will receive AX-158 treatment for 28 days with a 30 day safety follow-up period.
  Arms: AX-158 - (Arm 1)
Drug: Placebo — Subjects randomized to this arm will receive placebo treatment for 28 days with a 30 day safety follow-up period.
  Arms: Placebo - (Arm 2)

SUMMARY:
Proof of concept study to assess the safety and tolerability of AX-158 in patients with mild to moderate psoriasis. Patients will be evaluated for a 28-day treatment period with either AX-158 or Placebo and then followed for an additional 30 days for safety.

DETAILED DESCRIPTION:
This is a Phase 2a Proof of Concept randomized, double-blind, placebo-controlled study to investigate the safety and tolerability of AX-158 in patients with mild to moderate Psoriasis. Participants will be randomized 2:1 to receive AX-158 or Placebo. A total of 30 participants will be treated for 28 days and followed for an additional 30 days for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to provide informed consent and able to comply with the study procedures and restrictions.
2. Diagnosis of plaque psoriasis for ≥3 months at time of screening.
3. Male or female subjects age 18 to 60 years, inclusive, at the time of informed consent.
4. Body mass index (BMI) 18 to 40 kg/m2, inclusive, where BMI (kg/m2) is calculated by body weight (kg)/height2 (m2).
5. Female subjects may be enroled if the following criteria are met:

   1. Documented to be surgically sterile or postmenopausal or practicing true abstinence for at least 28 days prior to investigational product (IP) administration until 30 days (duration of ovulatory cycle) after the last IP administration and having a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to the start of IP administration, or
   2. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to the start of IP administration.
   3. WOCBP must agree to follow instructions for methods of contraception as described in Appendix 18.2 for the duration of treatment with IP plus 5 half-lives of IP (50 hours) plus 30 days (duration of ovulatory cycle) after the last IP administration.
   4. Women must not be pregnant, lactating, breastfeeding, or planning pregnancy during the study period.
6. Male subjects who are sexually active with WOCBP may be enrolled if they are

   1. Documented to be surgically sterile (vasectomy), or
   2. Practicing true abstinence for 90 days after the last IP administration, or
   3. Males who are sexually active with WOCBP must agree to follow instructions for methods of contraception for the duration of treatment with IP plus 5 half-lives of the IP plus 90 days (duration of sperm turnover) after the last IP administration. In addition, male subjects must be willing to refrain from sperm donation during this time.
7. Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements and must still undergo pregnancy testing as described in inclusion criterion #6b.
8. Fully vaccinated for COVID-19 per local regulations and site standard of care (SOC).

Exclusion Criteria:

1. Diagnosis of non-plaque psoriasis (guttate, inverse, pustular, erythrodermic).
2. Diagnosis of psoriatic arthritis, uveitis, inflammatory bowel disease, or other immune-mediated conditions that are commonly associated with psoriasis for which a subject requires current systemic (oral, subcutaneous, or intravenous [IV]) (including corticosteroids, immunosuppressants, biologics) immunosuppressant medical treatment. Certain therapies such as non-steroidal anti-inflammatory drugs may be permitted at the discretion of the medical monitor.
3. Psoriasis affecting the scalp only.
4. Inability to tolerate oral medication.
5. A clinically significant history of gastrointestinal disorder likely to influence absorption of IP.
6. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular, or metabolic dysfunction.
7. Participation in a clinical study and/or receipt of an IP within the previous 3 months or 5 half-lives, whichever is longer, before administration of the first dose of IP.
8. History or evidence of active infection and/or febrile illness within 7 days of first administration of IP.
9. History of serious bacterial, fungal, or viral infections that required hospitalization and IV antibiotic treatment within 90 days prior to screening, or any recent serious infection requiring antibiotic treatment within 30 days of IP administration.
10. Has received a live vaccine within 60 days of first dose of IP.
11. Current clinical radiographic or laboratory evidence of active tuberculosis (TB), or any history of or significant risk for TB.
12. Any major surgery within 4 weeks of IP administration.
13. Has unstable cardiovascular disease, defined as a recent clinical deterioration (eg, unstable angina, rapid atrial fibrillation) in the last 3 months or a cardiac hospitalization within the last 3 months.
14. History of malignancy (solid organ or hematologic including myelodysplastic syndrome) or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell or squamous cell carcinoma that has been treated with no evidence of recurrence).
15. Has used topical medications/treatments that could affect psoriasis or sPGA evaluation (including, but not limited to, mild to moderate corticosteroids [eg, hydrocortisone cream, triamcinolone acetonide], calcineurin inhibitor, calcipotriol, salicylic acid/other keratolytic, coal tar, short contact dithranol) within 4 weeks of the first administration of IP.
16. Has received phototherapy that could affect psoriasis or sPGA evaluation (eg, narrowband ultraviolet B [UVB] psoralen [oral or topical] with local UVA) within 4 weeks of the first administration of IP.
17. Has received any systemic non-biologic medications/treatments (including, but not limited to, methotrexate, ciclosporin, acitretin, and apremilast) or any systemic biologic medications/treatments (including, but not limited to etanercept, efalizumab, infliximab, adalimumab, ustekinumab, secukinumab, and ixekizumab) that could affect psoriasis or sPGA evaluation within 4 weeks of the first administration of the IP.
18. Chest X-ray findings suspicious of infection at screening. Subjects may be rescreened and if deemed eligible may be randomized within 28 days of completing an appropriate course of antibiotic treatment for pulmonary infection. If a chest X-ray has been performed within 6 months of the screening visit and the report and results are available, then a chest X-ray is not required at the screening visit.
19. Clinically significant history of previous allergy and/or sensitivity to AX-158 or any of the excipients contained within AX-158.
20. Clinically significant abnormal test results for serum biochemistry, hematology, and/or urine analyses within 28 days prior to first dose administration of the IP:

    1. Leukopenia defined as absolute white blood cell count <3000/mm3 within 28 days of dosing with IP on Day 1.
    2. Lymphopenia defined as absolute lymphocyte count <500/mm3 within 28 days of dosing with IP on Day 1.
    3. Neutropenia defined as absolute neutrophil count <1000/mm3 within 28 days of dosing with IP on Day 1.
    4. Moderate to severe thrombocytopenia defined as platelet count <100,000/mm3 within 28 days of dosing with IP on Day 1.
    5. Moderate to severe anemia defined as hemoglobin <9 g/dL within 28 days of dosing with IP on Day 1.
    6. Total serum bilirubin, alkaline phosphatase, aspartate transaminase and alanine transaminase >1.5 × upper limit of normal (ULN). If total bilirubin is above the ULN and is then fractionated, direct bilirubin must be within normal limits.
21. Subject with a positive urinary drug screen (including alcohol and cotinine) test results, determined within 28 days before the first dose administration of the IP. A positive test result may be repeated at the investigator's discretion.
22. Clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 28 days before first dose of IP including a QRS >120 ms, PR interval >220 ms and QT interval corrected using Fredericia's formula >450 ms.
23. Clinically significant abnormalities in vital signs and physical examination determined within 28 days before first dose of IP.
24. Subjects with a positive COVID-19 test on admission per local regulations and site SOC.
25. Any other condition that, in the investigator's judgement, will substantially increase the risk to the subject if they participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | Baseline to 28 days of treatment
  The frequency of treatment-emergent adverse events (TEAEs) either started after initial treatment or intensified in severity

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) -25 | Baseline to 28 days of treatment
  Proportion of subjects receiving AX-158 compared to placebo with PASI 25
Psoriasis Area and Severity Index (PASI) -50 | Baseline to 28 days of treatment
  Proportion of subjects receiving AX-158 compared to placebo with PASI 50
Psoriasis Area and Severity Index (PASI) -75 | Baseline to 28 days of treatment
  Proportion of subjects receiving AX-158 compared to placebo with PASI 75
Psoriasis Area and Severity Index (PASI) - 100 | Baseline to 28 days of treatment
  Proportion of subjects receiving AX-158 compared to placebo with PASI 100
Biomarkers | Baseline to 28 days of treatment
  Change from baseline in histological markers of psoriasis in skin biopsies.
Static Physician Global Assessment (sPGA) | Baseline to 28 days of treatment
  Proportion of patients receiving AX-158 compared to placebo who achieve sPGA score of 0 or 1

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Accellacare Northamptonshire, Corby
  - Accellacare Warwickshire, Coventry
  - MEU, Manchester
  - Accellacare North London, Northwood
  - Accellacare South London, Orpington
  - Accellacare Yorkshire, Shipley

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borroto A, Reyes-Garau D, Jimenez MA, Carrasco E, Moreno B, Martinez-Pasamar S, Cortes JR, Perona A, Abia D, Blanco S, Fuentes M, Arellano I, Lobo J, Heidarieh H, Rueda J, Esteve P, Cibrian D, Martinez-Riano A, Mendoza P, Prieto C, Calleja E, Oeste CL, Orfao A, Fresno M, Sanchez-Madrid F, Alcami A, Bovolenta P, Martin P, Villoslada P, Morreale A, Messeguer A, Alarcon B. First-in-class inhibitor of the T cell receptor for the treatment of autoimmune diseases. Sci Transl Med. 2016 Dec 21;8(370):370ra184. doi: 10.1126/scitranslmed.aaf2140. PMID 28003549
- [Background] Roy E, Togbe D, Holdorf AD, Trubetskoy D, Nabti S, Kublbeck G, Klevenz A, Kopp-Schneider A, Leithauser F, Moller P, Bladt F, Hammerling G, Arnold B, Pawson T, Tafuri A. Nck adaptors are positive regulators of the size and sensitivity of the T-cell repertoire. Proc Natl Acad Sci U S A. 2010 Aug 31;107(35):15529-34. doi: 10.1073/pnas.1009743107. Epub 2010 Aug 13. PMID 20709959
- [Background] Roy E, Togbe D, Holdorf A, Trubetskoy D, Nabti S, Kublbeck G, Schmitt S, Kopp-Schneider A, Leithauser F, Moller P, Bladt F, Hammerling GJ, Arnold B, Pawson T, Tafuri A. Fine tuning of the threshold of T cell selection by the Nck adapters. J Immunol. 2010 Dec 15;185(12):7518-26. doi: 10.4049/jimmunol.1000008. Epub 2010 Nov 15. PMID 21078909
- [Background] Gil D, Schamel WW, Montoya M, Sanchez-Madrid F, Alarcon B. Recruitment of Nck by CD3 epsilon reveals a ligand-induced conformational change essential for T cell receptor signaling and synapse formation. Cell. 2002 Jun 28;109(7):901-12. doi: 10.1016/s0092-8674(02)00799-7. PMID 12110186
- [Background] Juraske C, Wipa P, Morath A, Hidalgo JV, Hartl FA, Raute K, Oberg HH, Wesch D, Fisch P, Minguet S, Pongcharoen S, Schamel WW. Anti-CD3 Fab Fragments Enhance Tumor Killing by Human gammadelta T Cells Independent of Nck Recruitment to the gammadelta T Cell Antigen Receptor. Front Immunol. 2018 Jul 9;9:1579. doi: 10.3389/fimmu.2018.01579. eCollection 2018. PMID 30038626
- [Background] Borroto A, Arellano I, Blanco R, Fuentes M, Orfao A, Dopfer EP, Prouza M, Suchanek M, Schamel WW, Alarcon B. Relevance of Nck-CD3 epsilon interaction for T cell activation in vivo. J Immunol. 2014 Mar 1;192(5):2042-53. doi: 10.4049/jimmunol.1203414. Epub 2014 Jan 27. PMID 24470497
- [Background] Borroto A, Arellano I, Dopfer EP, Prouza M, Suchanek M, Fuentes M, Orfao A, Schamel WW, Alarcon B. Nck recruitment to the TCR required for ZAP70 activation during thymic development. J Immunol. 2013 Feb 1;190(3):1103-12. doi: 10.4049/jimmunol.1202055. Epub 2012 Dec 24. PMID 23267019
- [Background] Lettau M, Pieper J, Gerneth A, Lengl-Janssen B, Voss M, Linkermann A, Schmidt H, Gelhaus C, Leippe M, Kabelitz D, Janssen O. The adapter protein Nck: role of individual SH3 and SH2 binding modules for protein interactions in T lymphocytes. Protein Sci. 2010 Apr;19(4):658-69. doi: 10.1002/pro.334. PMID 20082308
- [Background] Yiemwattana I, Ngoenkam J, Paensuwan P, Kriangkrai R, Chuenjitkuntaworn B, Pongcharoen S. Essential role of the adaptor protein Nck1 in Jurkat T cell activation and function. Clin Exp Immunol. 2012 Jan;167(1):99-107. doi: 10.1111/j.1365-2249.2011.04494.x. PMID 22132889